CLINICAL TRIAL: NCT03181204
Title: Modeling Bronchial Epithelia Modifications Associated With Chronic Obstructive Pulmonary Disease (COPD) Using Induced Pluripotent Stemcells (iPS)
Brief Title: Modeling Bronchial Epithelium Modifications Associated With COPD Using iPS
Acronym: INVECCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9791; 2017-A00252-51 (Other: RCB number)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — This study will general cell cultures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients likely to develop COPD: Patients in this group are relatively light smokers who have developed chronic obstructive lung disease (COPD).
  Intervention: Bronchial biopsy
  Intervention: Skin biopsy
  Intervention: Blood sample
  Interventions: Procedure: Bronchial biopsy; Procedure: Skin biopsy; Procedure: Blood sample
- Patients not likely to develop COPD: Patients in this group are heavy smokers who have no signs of chronic obstructive lung disease (COPD).
  Intervention: Bronchial biopsy
  Intervention: Skin biopsy
  Intervention: Blood sample
  Interventions: Procedure: Bronchial biopsy; Procedure: Skin biopsy; Procedure: Blood sample

INTERVENTIONS:
Procedure: Bronchial biopsy — The bronchial biopsy is part of this study's inclusion criteria and is required during routine care for the patient. Bronchial fibroscopy is performed under general or local anesthesia. Biopsies are performed using forceps and according to current recommendations. One biopsy will be fixed immediately in RCL2 medium while the others (between 3 and 6) will be kept in isotonic saline and rapidly prepared for air-liquid-interface (ALI) cell culture.
Procedure: Skin biopsy — The skin biopsy will be performed after local anesthesia by hypodermic injection of a 1% Xylocaine solution. A single sample of a skin fragment about 3 mm in diameter will be necessary.
Procedure: Blood sample — The blood sample will be taken at the end of the cutaneous biospy, approximately 20 ml of blood will be collected.

SUMMARY:
The primary objective of this study is to to verify the feasibility of obtaining and comparing two epithelia in two populations based on the following experiments:

* Differentiation of an Induced Pluripotent Stem cell (iPS) clone derived from cutaneous biopsy in a population of heavy smokers (plus patients with chronic obstructive pulmonary disease) in order to obtain differentiated bronchial epithelia in vitro.
* For each of these same patients, generation of bronchial epithelium in vitro from bronchial biopsy using human bronchial epithelial cells (HBECs) in air-liquid interface (ALI) cultures.

DETAILED DESCRIPTION:
Secondary objectives:

* Confrontation of the two models of in vitro generation of bronchial epithelium by iPS and ALI in order to validate our model of study of the human bronchial epithelium COPD generated by the iPS.
* Inducing a "COPD-like" epithelial phenotype by exposing the bronchial epithelia generated from the iPS to a source of in vitro toxin (tobacco) and studying its effects by transcriptomic analysis via high-throughput sequencing (NGS) at key steps during the model.
* Demonstrate the feasibility of obtaining iPS from peripheral blood sampling.

ELIGIBILITY:
Inclusion Criteria for COPD patients:

* The patient has given his/her signed, informed consent
* Forced expiratory volume in 1 second / forced vital capacity < 0.7 [FEV1/FVC < 0.7]
* FEV1 < 50% of predicted value
* Exclusion of other respiratory pathologies, based on anamnesis, computed tomography and complementary respiratory function tests and transthoracic ultrasound,
* Smoking >10 pack-years, ongoing or weaned
* Absence of exacerbation or intercurrent infectious episode for at least 4 weeks at time of inclusion
* Medical indication for a bronchial fibroscopy (indication validated by the physician in charge of the patient and the study investigating physician): pulmonary peripheral nodule exploration with computed tomography, interventional endoscopy for emphysema reduction, removal of foreign bodies, other indications.
* Absence of contraindications for bronchial biopsy (left to physician's discretion): not limited to: regular intake of anticoagulants or anti-platelet aggregation, hemostasis abnormalities

Inclusion Criteria for smokers:

* The patient has given his/her signed, informed consent
* Forced expiratory volume in 1 second / forced vital capacity > 0.7 [FEV1/FVC > 0.7]
* FEV1 > 80% of predicted value
* Exclusion of other respiratory pathologies, based on anamnesis, computed tomography (absence of extensive emphysema lesions defined by the presence of less than <5% relative surface area occupied by densities less than 910 UH (measured on millimeter cuts)) and respiratory function tests (Residual Volume <120%, Diffusion Capacity for Carbon Monoxide > 60% and Total Pulmonary Capacity> 120%) and transthoracic ultrasound (normal),
* Smoking >40 pack-years, ongoing or weaned
* Absence of exacerbation or intercurrent infectious episode for at least 4 weeks at time of inclusion
* Medical indication for a bronchial fibroscopy (indication validated by the physician in charge of the patient and the study investigating physician): pulmonary peripheral nodule exploration with computed tomography, interventional endoscopy for emphysema reduction, removal of foreign bodies, other indications.
* Absence of contraindications for bronchial biopsy (left to physician's discretion): not limited to: regular intake of anticoagulants or anti-platelet aggregation, hemostasis abnormalities

Exclusion Criteria:

* Contra-indication for bronchial fibroscopy and cutaneous biopsy
* Deficiency in α-1 antitrypsin
* Significant bronchiectasis on chest computed tomography scan
* Colonization of the airways by Pseudomonas Aeroginosa or Aspergillus
* Chemotherapy or other cytotoxic treatments in the last 12 months
* Systemic corticotherapy in the 4 weeks prior to inclusion
* Long-term antibiotic treatment, notably by macrolides
* Any other treatment that may affect the bronchial epithelium, this being left to the discretion of the investigating physician
* Consumer of illicit drugs or alcohol
* Participant in an exclusion period determined by a previous study
* Subject not affiliated with, or not beneficiary of, a social security plan.
* Pregnant or nursing women according to Article L1121-5 of the Public Health Code.
* Vulnerable persons according to Article L1121-6 of the Public Health Code
* An adult who is protected or incapable of giving consent in accordance with Article L1121-8 of the Public Health Code
* Subject deprived of freedom by judicial or administrative decision.
* Those patients for whom two epithelia cultures (1 from bronchial biopsy ("ALI") and 1 from fibroblast reprogrammation of redifferentiated iPS ("iALI")) were not obtained will be excluded (post-inclusion).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study includes patients with chronic obstructive pulmonary disease, as well as patients without chronic obstructive pulmonary disease, but who are heavy smokers.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
functional bronchial epithelium from iPS? | Day 0 + culture (cross-sectional study)
  Was a functional bronchial epithelium obtained from the patient's induced pluripotent stem cells from blood or fibroblasts? (yes/no)
functional bronchial epithelium from HBEC-ALI? | Day 0 + culture (cross-sectional study)
  Was a functional bronchial epithelium obtained from the patient's bronchial biopsy: human bronchial epithelial cell culture on an air-liquid-interface? (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Centre Hospitalier Universitaire de Montpellier, Montpellier, France

REFERENCES:
- [Result] Ahmed E, Fieldes M, Mianne J, Bourguignon C, Nasri A, Vachier I, Assou S, Bourdin A, De Vos J. Generation of four severe early-onset chronic obstructive pulmonary disease (COPD) patient-derived induced pluripotent stem cell lines from peripheral blood mononuclear cells. Stem Cell Res. 2021 Oct;56:102550. doi: 10.1016/j.scr.2021.102550. Epub 2021 Sep 27. PMID 34624616
- [Result] Fieldes M, Ahmed E, Bourguignon C, Mianne J, Vernisse C, Fort A, Vachier I, Bourdin A, Assou S, De Vos J. [Modelling the bronchial epithelium in chronic obstructive pulmonary disease using human induced pluripotential stem cells]. Rev Mal Respir. 2020 Mar;37(3):197-200. doi: 10.1016/j.rmr.2020.02.003. Epub 2020 Mar 4. French. PMID 32146059
- See also: INVECCO on the Open Science Framework — http://osf.io/vhtak